CLINICAL TRIAL: NCT04172220
Title: Variation of the Neutrophil To Lymphocyte Ratio During Opioid-Free General Anesthesia Associated With Thoracic Wall Blocks Vs General Anesthesia, in Breast Cancer Quadrantectomy: a Randomized Controlled Trial
Brief Title: Does Type of Anesthesia Influence Inflammation Change After Breast Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CRO-2019-26
Record Dates: First submitted 2019-11-14; First posted 2019-11-21 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Female
Keywords: Breast Cancer; PECS; Neutrophil to Lymphocyte ratio; Quadrantectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Midazolam; Anesthesia, General

STUDY DESIGN:
Intervention Model Description: Single center, open label randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS + Opioid-free GA (Experimental): Loco-regional anesthesia with PEC I and serratus plane block with an echoguided technique and opioid-free general anesthesia
  Interventions: Drug: Midazolam; Procedure: PECS; Procedure: Opioid-free general anesthesia; Procedure: Postoperative analgesia
- GA (Active Comparator): General anesthesia
  Interventions: Drug: Midazolam; Procedure: General anesthesia; Procedure: Postoperative analgesia

INTERVENTIONS:
Drug: Midazolam — 1-2 mg of Midazolam as premedication.
Procedure: PECS — Loco-regional anesthesia: PEC I and serratus plane block with an echoguided technique.
  For the PEC I: infiltration of 10 ml of local anesthetic (Levobupivacaine 0.25% or Ropivacaine 0.5%) between the bands of the pectoralis major muscle and the small pectoralis muscle at the height of the third rib on the anterior axillary line.
  For the serratus plane block: identification of the fifth rib on the average axillary line and infusion of about 20 ml of local anesthetic (Levobupivacaine 0.25% or Ropivacaine 0.5%) between the bands of large dorsal muscle and of the anterior serratus muscle.
  Arms: PECS + Opioid-free GA
Procedure: Opioid-free general anesthesia — Induction with Propofol 1.5-2 mg/kg; laryngeal mask for airway management after eventual administration of Rocuronium 0.6 mg/kg. Anesthesia will be maintained with Propofol in Target-Controlled Infusion (TCI) of 6 mcg/ml, subsequently modified to maintain a Bispectral Index (BIS) value between 40 and 60.
  Fentanyl 50ug in bolus IV, in case of mean arterial pressure or heart rate increase >20%.
  In case of hypotension: 5mg ephedrine and infusion of 250 ml Lactated Ringer.
  Arms: PECS + Opioid-free GA
Procedure: General anesthesia — Induction with Propofol 1.5-2 mg/kg; Fentanyl 1μg/kg; laryngeal mask for airway management after eventual administration of Rocuronium 0.6 mg/kg. Anesthesia will be maintained with Propofol in TCI of 6 mcg/ml, subsequently modified to maintain a BIS value between 40 and 60.
  Fentanyl 50ug in bolus IV, in case of mean arterial pressure or heart rate increase >20%.
  In case of hypotension: 5mg ephedrine and infusion of 250 ml Lactated Ringer.
  Arms: GA
Procedure: Postoperative analgesia — Paracetamol 1000 mg every 8 hours for the first 24 hours, Ketorolac 30 mg in case of pain control failure (Numeric Rating Scale- NRS>4) which can be administered every 8 hours at most (max 90 mg / 24 hours), Morphine 10-20 mg IV in 24 hours as rescue analgesia.

SUMMARY:
The Neutrophil to Lymphocyte Ratio (NLR) is a frequently used biomarker of the systemic inflammatory response and is considered one of the most sensitive markers of inflammation. Many studies have documented the association between the use of opioid drugs in the acute phase -as it can be considered the use during general anesthesia- and the increase of the NLR value. Such increase could determine a temporary phase of immunodepression in the immediate post operative period with consequent increase of the inflammatory state.

This study intends to assess whether different anesthetic techniques can be associated with different variations of the intra-patient NLR value between pre- and post-surgery. Patient will be randomized to receive either local regional anesthesia protocols with thoracic wall blocks (PEC I and serratus plane block) associated with opioid-free general anesthesia (PECS + Opioid-free GA) or general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* First diagnosis of histologically confirmed breast cancer
* Candidate to external quadrantectomy and axillary surgery (biopsy of the sentinel lymph node and possible axillary lymphadenectomy)
* Able to provide adequate informed consent
* With intact cognitive abilities

Exclusion Criteria:

* Ongoing pregnancy
* In therapy or in follow-up for other cancers at the time of the study
* Concurrent therapy with opioids or other drugs, for chronic pain conditions related to cancer or other diseases
* History of documented allergy or previous adverse reaction to local anesthetics
* Documented history of anesthesiology related problems during previous surgical interventions or history of problems in airway management
* Unable to comply to study protocol schedule for logistic or other reasons
* Refusal to participate to the study (absence of signed informed consent)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
24h NLR variation | Pre-operative and at 24 hours after the end of surgery
  Intra-patient variation of the NLR value between the pre-operative and the first post-operative day

SECONDARY OUTCOMES:
1h NLR variation | Pre-operative, 1 hour and 24 hours after the end of surgery
  Intra-patient variation of the NLR value between pre-operative and 1 hour after the end of surgery, and between 1 hour after the end of surgery and 24 hours after the end of surgery
Opioid consumption | 24 hours
  Consumption of intra-operative Fentanyl and post-operative Morphine hydrochloride during the first 24 hours after surgery
Complication | until hospital discharge, an average of 48 hours
  Complications related to the loco-regional anesthesia technique or to the administration of the local anesthetic. For pain evaluation, the validated Numeric Rating Scale (NRS) will be used, the score ranges from 0 to 10 with higher values corresponding to worse pain.
Chronic pain | 3, 6 and 12 months after surgery
  Chronic pain after surgery will be assessed with Brief Pain Inventory questionnaire (composed by pain severity and pain interference scores). "Douleur Neuropathique 4" (DN4) questionnaire will be used for the identification of neuropathic pain. All the scores range from 0 to 10, with 10 indicating the worst results.
Change in the levels of circulating cytokines in the post-operative period (one hour and 24 hours after surgery), compared to the baseline pre-operative values, in the two arms | 24 hours
  differences in fold change of selected cytokines between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Brescia, MD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO), IRCCS
Locations (1):
- Centro di Riferimento Oncologico di Aviano (CRO), IRCCS, Aviano, PN, Italy

REFERENCES:
- [Derived] Brescia F, Favero A, Segatto I, Massarut S, Zanier C, Fabiani F, Nadalini E, Morabito A, Montico M, Zucchetto A, Zanussi S, Baldassarre G, Belletti B. Impact of opioid-free general anesthesia with locoregional blocks during breast cancer surgery on systemic inflammatory response: results from a randomized controlled trial. Reg Anesth Pain Med. 2025 Jun 25:rapm-2025-106504. doi: 10.1136/rapm-2025-106504. Online ahead of print. PMID 40562448